CLINICAL TRIAL: NCT06004492
Title: Effectiveness of an Integrated Program Combining Technology-assisted Blended Learning in Enhancing Motivational Interviewing Knowledge, Skills, Self-efficacy, and Its Impact on Patient Medication Adherence
Brief Title: Technology-assisted Blended Learning on Motivational Interviewing for Mental Health Nurses and Its Clinical Impact
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Responsible Party: Principal Investigator, Wen I Liu, Distinguished Professor, National Taipei University of Nursing and Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: blended learning
Record Dates: First submitted 2023-08-16; First posted 2023-08-22 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Nurse's Role
Keywords: blend learning; technology-assisted practice learning; motivational interviewing; mentaj health nurse

STUDY DESIGN:
Intervention Model Description: blended learning program (8 hours of workshops and four months of practical learning on technology platforms); control group received conventional education
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- blended learning program (Placebo Comparator): 8 hours of workshops and four months of practical learning on technology platforms
  Interventions: Behavioral: blended learning program
- conventional education (No Intervention): conventional education

INTERVENTIONS:
Behavioral: blended learning program — blended learning program: 8 hours of workshops and four months of practical learning on technology platforms.
  Other Names: Motivational Interviewing Care Competence Based on Blended Learning
  Arms: blended learning program

SUMMARY:
Medication adherence is the primary care to stabilize the symptoms of patients with schizophrenia, but more than half of community patients still do not adhere to medication. According to the latest research of our team, the motivational interviewing may be more effective in promoting medication adherence than the insight. In the past, there was a lack of theoretical and empirical motivational interviewing and integrated medication adherence program. Therefore, the first year of this plan has completed the construction of integrated medication adherence. Considering the current lack of training and promotion of the blended learning model assisted by convenient and effective mobile technology.

Aim: To develop and evaluate the effectiveness of an integrated program combining technology-assisted blended learning on motivational interviewing knowledge, skills, and self-efficacy for psychiatric mental health nurses, and its clinical impact.

ELIGIBILITY:
Inclusion Criteria:

* mental health registered Nurse who take care of patients.

Exclusion Criteria:

* expected to leave the job within two months
* over 65 years old

Max Age: 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 274 (Actual)
Dates: Start 2022-09-08 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
motivational interviewing skill | The time points of measurement are the baseline for nurses, the changes 8 hours after the workshop training, and the changes 4 months after the technology-assisted learning.
  Motivational Interviewing skill is a 12-items assessment tool.Total scores is range between 0 and 12, with a higher score indicating better skill.

SECONDARY OUTCOMES:
Motivational Interviewing Knowledge and Attitudes Test (MIKAT) | The time points of measurement are the baseline for nurses, the changes 8 hours after the workshop training, and the changes 4 months after the technology-assisted learning.
  Motivational Interviewing Knowledge and Attitudes Test is a 29-items self-reporting scales.Total scores on the MIKAT range between 0 and 29, with a higher score indicating better knowledge.
Motivational Interviewing Confidence Survey (MICS) | The time points of measurement are the baseline for nurses, the changes 8 hours after the workshop training, and the changes 4 months after the technology-assisted learning.
  MICS is a 24-items self-reporting with 10-point Likert scale.Total scores on the MICS range between 0 and 240, with a higher score indicating better self-efficacy.
Medication Adherence Rating Scale (MARS) | The time points of measurement are the baseline for patients, the changes 6 months after motivational interviewing care based on blended learning, and the changes at 9 months in clinical effects.
  The Medication Adherence Rating Scale(MARS) is a 10-item self-reporting multidimensional instrument describing three dimensions: medication adherence behavior (items 1-4), attitude toward taking medication (items 5-8) and negative side effects and attitudes to psychotropic medication (items 9-10). sponse consistent with non-adherence is coded as 0, whereas a response consistent with adherence is coded as 1. For questions 1-6 and 9-10, a no response is indicative of adherence and is coded as 1, while for questions 7 and 8, a yes response is indicative of adherence and is coded as 1. Total scores on the MARS may range between 0 and 10, with a higher score indicating better medication adherence.
Drug Attitude Inventory (DAI-10) | The time points of measurement are the baseline for patients, the changes 6 months after motivational interviewing care based on blended learning, and the changes at 9 months in clinical effects.
  The Drug Attitude Inventory(DAI-10) contains six items that a patient who is fully adherent to prescribed medication would answer as 'True', and four they would rate as 'False'. Scores are allocated to each answer and the total score is calculated in the same way as for the DAI-30. The range is -4 to 6 points. The higher the score, the more positive the attitude of taking the medicine, with 0 points as the cut-off point, above 0 means the attitude of taking the medicine is positive; below 0 means the attitude of taking the medicine is negative
University of Rhode Island Changed Assessment (URICA) | The time points of measurement are the baseline for patients, the changes 6 months after motivational interviewing care based on blended learning, and the changes at 9 months in clinical effects.
  The University of Rhode Island Change Assessment Scale (URICA) is a 32 item self-report measure that includes 4 subscales measuring the stages of change: Precontemplation, Contemplation, Action, and Maintenance (there is also a 24 item version). Responses are given on a 5 point Likert scale ranging from (1=strong disagreement to 5=strong agreement),Calculate the score with its calculation formula, and get a score ranging from -2 to 14. The higher the score, the stronger the motivation to change.
Brief Psychiatric Rating scale (BPRS) | The time points of measurement are the baseline for patients, the changes 6 months after motivational interviewing care based on blended learning, and the changes at 9 months in clinical effects.
  The Brief Psychiatric Rating scale(BPRS) assesses the level of 18 symptom constructs such as hostility, suspiciousness, hallucination, and grandiosity. It is particularly useful in gauging the efficacy of treatment in patients who have moderate to severe psychoses.Total scores on the MARS may range between 0 and 10, with a higher score indicating better medication adherence.This scale is scored from 0-6, with a total of 16 items, and the total score ranges from 0 to 96. The higher the score, the more obvious the psychiatric symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- National Taipei University of Nursing and Health Sciences, Taipei, Taiwan